CLINICAL TRIAL: NCT01478048
Title: A Phase 2, Randomized Study of Bortezomib/Dexamethasone With or Without Elotuzumab in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Bortezomib and Dexamethasone With or Without Elotuzumab to Treat Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA204-009; 2011-002695-16 (EudraCT Number)
Record Dates: First submitted 2011-11-02; First posted 2011-11-23 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Elotuzumab + Bortezomib + Dexamethasone (Experimental): On days of Elotuzumab infusion: Dexamethasone (8mg IV + 8mg Oral) will be administered other days Dexamethasone 20 mg Oral will be administered
  Interventions: Biological: Elotuzumab; Drug: Bortezomib; Drug: Dexamethasone
- Arm B: Bortezomib + Dexamethasone (Active Comparator)
  Interventions: Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Biological: Elotuzumab — Solution; Intravenous (IV); 10 mg/kg; (Cycles 1 & 2: Days 1, 8 & 15; Cycles 3-8: Days 1 & 11; Cycle 9+: Days 1 & 15); Until subject meets criteria for discontinuation of study drug
  Other Names: BMS-901608
  Arms: Arm A: Elotuzumab + Bortezomib + Dexamethasone
Drug: Bortezomib — Solution; IV; 1.3 mg/m2; (Cycles 1 - 8: Days 1, 4, 8, 11; Cycles 9+: Days 1, 8, 15); Until subject meets criteria for discontinuation of study drug
  Other Names: Velcade®
Drug: Dexamethasone — Tablets; Oral; 20 mg; (Cycles 1& 2: once daily on Days 2, 4, 5, 8, 9, 11; Cycles 3-8: once daily on Days 2, 4, 5, 9, 12; Cycles 9+: once daily on Days 2, 8, 9, 16); Until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Intensol®; Dexpak®; Taperpak®
  Arms: Arm A: Elotuzumab + Bortezomib + Dexamethasone
Drug: Dexamethasone — Tablets; Oral; 8 mg; (Cycles 1& 2: Days 1, 8, 15; Cycles 3-8: Days 1 &11; Cycles 9+; Days 1 & 15); Until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Intensol®; Dexpak®; Taperpak®
  Arms: Arm A: Elotuzumab + Bortezomib + Dexamethasone
Drug: Dexamethasone — Solution; IV; 8 mg; (Cycles 1& 2: Days 1, 8, 15; Cycles 3-8: Days 1 &11; Cycles 9+; Days 1 & 15); Until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Intensol®; Dexpak®; Taperpak®
  Arms: Arm A: Elotuzumab + Bortezomib + Dexamethasone
Drug: Dexamethasone — Tablets; Oral; 20 mg; (Cycles 1-8 once daily on Days 1, 2, 4, 5, 8, 9, 11, 12; Cycles 9+ once daily on Days 1, 2, 8, 9, 15, 16); Until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Intensol®; Dexpak®; Taperpak®
  Arms: Arm B: Bortezomib + Dexamethasone

SUMMARY:
The purpose of the study is to determine whether the addition of Elotuzumab to Bortezomib/ Dexamethasone will prolong the time before myeloma worsens [progression free survival (PFS)].

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* Documented progression from most recent line of therapy
* Measurable disease
* 1 to 3 prior lines of therapy

  * Subjects may be proteasome inhibitor naive or have received prior proteasome inhibitor therapy provided all the following criteria are met:

    1. The subject did not discontinue any proteasome inhibitor due to intolerance or grade ≥ 3 toxicity
    2. The subject is not refractory to any proteasome inhibitor, defined as progression during treatment or within 60 days after the last dose
    3. The subject previously achieved a partial response (PR) or better to previous proteasome inhibitor (PI)

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance (MGUS), smoldering myeloma, or Waldenstrom's macroglobulinemia
* Active plasma cell leukemia
* Known Human immunodeficiency virus (HIV) infection or active hepatitis A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (75):
- United States (42):
  - Compassionate Cancer Res Grp, Corona, California
  - Local Institution, Corona, California
  - Local Institution, Long Beach, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Ucla Department Of Medicine, Los Angeles, California
  - Medical Oncology Care Associates, Orange, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Local Institution, Vallejo, California
  - Cancer Specialists of North FL, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Kaiser Permanente-Moanalua Medical Center, Honolulu, Hawaii
  - University Of Chicago Medical Center, Chicago, Illinois
  - Local Institution, Decatur, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Local Institution, Urbana, Illinois
  - Investigative Clinical Research Of Indiana, Llc, Indianapolis, Indiana
  - Local Institution, Hazard, Kentucky
  - University Of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Pikeville Medical Center Leonard Lawson Cancer Center, Pikeville, Kentucky
  - Cancer Center Of Acadiana, Lafayette, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mercy Medical Research Institute, Springfield, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Waverly Hematology Oncology, Cary, North Carolina
  - St. Agnes Hospital, Baltimore, Pennsylvania
  - Cancer Care Associates, Bethlehem, Pennsylvania
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Penn State Hershey Cancer Inst, Hershey, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Medical University Of South Carolina, Charleston, South Carolina
  - Local Institution, Greenville, South Carolina
  - Charles A. Sammons Cancer Center, Dallas, Texas
  - Northwest Cancer Center, Houston, Texas
  - Local Institution, Fairfax, Virginia
  - Local Institution, Seattle, Washington
- Local Institution, Halifax, Nova Scotia, Canada
- France (7):
  - Local Institution, Grenoble
  - Local Institution, Le Mans
  - Local Institution, Lille
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
- Italy (17):
  - Local Institution, Milan, Parma
  - Local Institution, Roma, Parma
  - Local Institution, Ancona
  - Local Institution, Bari
  - Local Institution, Bologna
  - Local Institution, Brescia
  - Local Institution, Florence
  - Local Institution, Genova
  - Local Institution, Lecce
  - Local Institution, Meldola (fc)
  - Local Institution, Modena
  - Local Institution, Pescara
  - Local Institution, Ravenna
  - Local Institution, Rimini
  - Local Institution, Roma
  - Local Institution, Rome
  - Local Institution, Torino
- Spain (8):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Murcia
  - Local Institution, Salamanca
  - Local Institution, Santiago Compostela
  - Local Institution, Toledo
  - Local Institution, Valencia
  - Local Institution, Zaragoza

REFERENCES:
- [Derived] Jakubowiak A, Offidani M, Pegourie B, De La Rubia J, Garderet L, Laribi K, Bosi A, Marasca R, Laubach J, Mohrbacher A, Carella AM, Singhal AK, Tsao LC, Lynch M, Bleickardt E, Jou YM, Robbins M, Palumbo A. Randomized phase 2 study: elotuzumab plus bortezomib/dexamethasone vs bortezomib/dexamethasone for relapsed/refractory MM. Blood. 2016 Jun 9;127(23):2833-40. doi: 10.1182/blood-2016-01-694604. Epub 2016 Apr 18. PMID 27091875
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 185 participants were enrolled, 152 participants were randomized. Reasons not randomized: 23 no longer met study criteria, 5 withdrew consent, 2 died, 3 had poor/non-compliance. 150 were treated with study drug. 2 participants were not treated: 1 withdrawal by subject and 1 physician decision.
Groups:
- Elotuzumab + Bortezomib + Dexamethasone: Elotuzumab: Solution; Intravenous (IV); 10 mg/kg; (Cycles 1 & 2: Days 1, 8 & 15; Cycles 3-8: Days 1 & 11; Cycle 9+: Days 1 & 15); Until participant meets criteria for discontinuation of drug Bortezomib: Solution; IV; 1.3 mg/m^2; (Cycles 1 - 8: Days 1, 4, 8, 11; Cycles 9+: Days 1, 8, 15); Until criteria met for discontinuation of drug. Days of Elotuzumab infusion: Dexamethasone (8mg IV + 8mg Oral) administered. Other days Dexamethasone 20 mg Oral administered Dexamethasone: Tablets; 20 mg; (Cycles 1& 2: once daily on Days 2, 4, 5, 8, 9, 11; Cycles 3-8: once daily on Days 2, 4, 5, 9, 12; Cycles 9+: once daily on Days 2, 8, 9, 16); Until criteria met for discontinuation. Dexamethasone: Tablets; 8 mg; (Cycles 1& 2: Days 1, 8, 15; Cycles 3-8: Days 1 &11; Cycles 9+; Days 1 & 15); Until criteria met for discontinuation of drug. Dexamethasone: Solution; IV; 8 mg; (Cycles 1& 2: Days 1, 8, 15; Cycles 3-8: Days 1 &11; Cycles 9+; Days 1 & 15); Until criteria met for discontinuation
- Bortezomib + Dexamethasone: Bortezomib: Solution; IV; 1.3 mg/m^2; (Cycles 1 - 8: Days 1, 4, 8, 11; Cycles 9+: Days 1, 8, 15); Until criteria met for discontinuation of study drug. Dexamethasone: Tablets; 20 mg; (Cycles 1-8 once daily on Days 1, 2, 4, 5, 8, 9, 11, 12; Cycles 9+ once daily on Days 1, 2, 8, 9, 15, 16); Until criteria is met for discontinuation of study drug
Period: Overall Study
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone
Started | 77 | 75
Received Treatment | 76 (1 randomized to E-Bd but received Bd. Included in E-Bd group for efficacy and Bd group for safety) | 74 (1 randomized to E-Bd but received Bd. Included in E-Bd group for efficacy and Bd group for safety)
Completed (Completed = Still on treatment) | 0 | 0
Not Completed | 77 | 75
Not completed — Disease Progression | 52 | 35
Not completed — study drug toxicity | 11 | 14
Not completed — Adverse Event | 2 | 11
Not completed — subject request to discontinue treatment | 3 | 5
Not completed — Withdrawal by Subject | 2 | 5
Not completed — non-specified | 6 | 4
Not completed — poor/non-compliance | 0 | 1
Not completed — no longer meets study criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who were randomized to a treatment arm were summarized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.48) | 65.1 (10.34) | 65.3 (9.88)
Age, Customized [Count of Participants; unit: Participants] — Less than (<); Greater than, equal to (≥).
  Participants
    < 65 years | 34 | 33 | 67
    ≥65 and <75 years | 28 | 28 | 56
    >= 75 years | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 42 | 37 | 79
Region of Enrollment [Count of Participants; unit: Participants] — Number of participants enrolled, by country, were summarized.
  Participants
    United States | 25 | 23 | 48
    Italy | 34 | 32 | 66
    France | 10 | 11 | 21
    Spain | 8 | 9 | 17
Prior Protease Inhibitor Use [Count of Participants; unit: Participants] — Categories presented as they were at randomization based on information collected via the Interactive Voice Recognition System (IVRS) system.
  Participants
    Yes | 38 | 37 | 75
    No | 39 | 38 | 77
Presence of At Least 1 FcγRIIIa V allele [Count of Participants; unit: Participants] — An allele is any one of a series of 2 or more different genes that may be on a specific chromosome. Categories presented as they were at randomization based on information collected via the Interactive Voice Recognition System (IVRS) system.
  Participants
    Yes | 55 | 54 | 109
    No | 22 | 21 | 43
Number of Prior Lines of Therapy [Count of Participants; unit: Participants] — Categories presented as they were at randomization based on information collected via the Interactive Voice Recognition System (IVRS) system.
  Participants
    1 line of prior therapy | 55 | 51 | 106
    2 or 3 lines of prior therapy | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Median Investigator-Assessed Progression-free Survival (PFS) Time (Months) From Randomization to Date of First Tumor Progression or Death Due to Any Cause - Randomized Participants
Description: PE was planned for after at least 103 events; it was analyzed after 111 events. Response was assessed: Day 1 (± 7 days) of each cycle per modified International Myeloma Working Group (IMWG) criteria; assessed using adequate tumor assessment (ATA) (ie, serum and urine M-protein tests performed within 14 days of each other; imaging if baseline measurable extramedullary plasmacytoma existed). Progression: Any of following: Increase of 25% from lowest response in 1 or more: serum and/or urine M-component; in those without measurable serum and urine M-protein levels, difference between involved and uninvolved free light chain (FLC) levels (absolute increase > 100 mg/L); Bone marrow plasma cell percentage (≥10%). Definite new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing lesions or plasmacytomas. Development of hypercalcemia attributed solely to the plasma cell proliferative disorder.
Time Frame: Randomization until 111 events (disease progression or death), up to May 2014, approximately 2 years
Population: Intent to treat (ITT), all randomized participants were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone
Number analyzed (Participants) | 77 | 75
Months | 9.7 [7.4 to 12.2] | 6.9 [5.1 to 10.2]
Statistical Analysis 1: Comparison: Elotuzumab + Bortezomib + Dexamethasone vs Bortezomib + Dexamethasone; Test type: Superiority or Other; p = 0.0923, Log Rank — Log Rank test was stratified by prior proteasome inhibitor use (Yes versus No), presence of at least 1 FcγRIIIa V allele (Yes versus No) and number of prior lines of therapy (1 versus 2 or 3) at randomization; Adjusted alpha level= 0.30; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.49 to 1.06]

2. Primary Outcome: Number of Investigator-Assessed Progression-free Survival Events From Randomization to Date of First Tumor Progression or Death Due to Any Cause - All Randomized Participants
Description: PE planned for after at least 103 events (progression/death); analyzed at 111 events. Those who neither progressed nor died were censored on the date of last adequate tumor assessment (ATA), which requires both serum and urine M-protein tests. If no post-baseline tumor assessments/no death, then censored on randomization day. Response assessed: Day 1 (± 7 days) each cycle; 30 and 60 days post treatment. Modified IMWG criteria used. Progression: Any of following: Increase of 25% in serum and/or urine M-component; if no measurable serum, urine M-protein levels, then difference between involved and uninvolved free light chain (FLC) levels (absolute increase > 100 mg/L) ; Bone marrow plasma cell percentage (≥10%). New bone lesions or soft tissue plasmacytomas or increase in size of existing lesions, plasmacytomas. Development of hypercalcemia attributed solely to plasma cell proliferative disorder. First dose occurs within 3 days of randomization.
Time Frame: Randomization until 111 events, up to May 2014, approximately 2 years
Population: Intent to treat (ITT), all randomized participants were analyzed.
Measure: Number; unit: Events (progression or death)
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone
Number analyzed (Participants) | 77 | 75
Events (progression or death) | 52 | 59

3. Secondary Outcome: Median Progression-free Survival Time (Months) From Randomization to Date of First Tumor Progression or Death Due to Any Cause, in Randomized Participants With at Least One FcγRIIIa V Allele
Description: PE was planned for after at least 103 events; it was analyzed after 111 events. Response was assessed: Day 1 (± 7 days) of each cycle per modified IMWG criteria; assessed using adequate tumor assessment (ATA) (ie, serum and urine M-protein tests performed within 14 days of each other; imaging if baseline measurable extramedullary plasmacytoma existed). Progression: Any of following: Increase of 25% from lowest response in 1 or more: serum and/or urine M-component; in those without measurable serum and urine M-protein levels, difference between involved and uninvolved FLC levels (absolute increase > 100 mg/L); Bone marrow plasma cell percentage (≥10%). Definite new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing lesions or plasmacytomas. Development of hypercalcemia attributed solely to the plasma cell proliferative disorder. Randomized participants with at least 1 FcγRIIIa V allele were a sub-set of all randomized participants.
Time Frame: Randomization until 111 events, up to May 2014, approximately 2 years
Population: All randomized participants who had at least one FcγRIIIa V allele were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone
Number analyzed (Participants) | 55 | 54
Months | 9.9 [6.1 to 13.9] | 8.1 [5.0 to 11.1]

4. Secondary Outcome: Investigator-Assessed Objective Response Rate (ORR) - All Randomized Participants
Description: ORR was calculated for participants with a best overall response (BOR) of partial response (PR) or better, including stringent complete response (sCR), complete response (CR), and very good partial response (VGPR). BOR was determined by the investigator based on myeloma tumor assessments using IMWG criteria: CR=Negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas, and < 5% plasma cells in bone marrow; sCR= CR + normal FLC ratio and absence of clonal cells in bone marrow; VGPR=Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein level + urine M-protein level < 100 mg per 24 hour; PR= ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hour. ORR= number of participants responding divided by total number of participants randomized, measured as a percentage.
Time Frame: Randomization until 111 events, up to May 2014, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone
Number analyzed (Participants) | 77 | 75
percentage of participants | 64.9 [53.2 to 75.5] | 62.7 [50.7 to 73.6]
Statistical Analysis 1: Comparison: Elotuzumab + Bortezomib + Dexamethasone vs Bortezomib + Dexamethasone; Test type: Superiority or Other; Difference using Chan-Zhang method = 2.3, 95% CI 2-sided [-13.2 to 17.8]

5. Primary Outcome: 1 Year Progression-Free Survival Rate - Randomized Participants
Description: PFS rate=Percentage probability of participants experiencing no progression or death up to 1 year, estimated using the Kaplan-Meier method. Response assessed by the investigator: Day 1 (± 7 days) of each cycle per modified IMWG criteria; assessed using ATA (ie, serum and urine M-protein tests performed within 14 days of each other; imaging done if baseline measurable extramedullary plasmacytoma existed). Progression: Any of the following: Increase of 25% from lowest response in 1 or more: serum and/or urine M-component; in those without measurable serum and urine M-protein levels, difference between involved and uninvolved FLC levels (absolute increase > 100 mg/L) ; Bone marrow plasma cell percentage (≥10%). Definite new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing lesions or plasmacytomas. Development of hypercalcemia attributed solely to the plasma cell proliferative disorder.
Time Frame: Year 1 after last participant was randomized
Population: All randomized participants were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone
Number analyzed (Participants) | 77 | 75
percentage probability | 0.39 [0.28 to 0.50] | 0.33 [0.22 to 0.44]

6. Secondary Outcome: Investigator-Assessed Objective Response Rate in Randomized Participants With at Least One FcγRIIIa V Allele
Description: ORR was calculated for participants with a BOR of PR or better, sCR, CR, and VGPR. BOR was determined by the investigator based on myeloma tumor assessments using IMWG criteria: CR=Negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas, and < 5% plasma cells in bone marrow; sCR= CR + normal FLC ratio and absence of clonal cells in bone marrow; VGPR=Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein level + urine M-protein level < 100 mg per 24 hour; PR= ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hour. ORR= number of participants responding divided by total number of participants randomized, measured as a percentage. Randomized participants with at least 1 FcγRIIIa V allele were a sub-set of all randomized participants.
Time Frame: Randomization until 111 events, up to May 2014, approximately 2 years
Population: All randomized participants who had at least one FcγRIIIa V allele at randomization were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone
Number analyzed (Participants) | 55 | 54
percentage of participants | 60.0 [45.9 to 73.0] | 61.1 [46.9 to 74.1]

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 60 days (assessed up to April 2017, approximately 63 months)
Arm/Group | Elotuzumab + Bortezomib + Dexamethasone | Bortezomib + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 37/75 | 39/75
Serious Adverse Events (participants affected / at risk) | 39/75 | 31/75
Other Adverse Events (participants affected / at risk) | 72/75 | 71/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab + Bortezomib + Dexamethasone (N=75) | Bortezomib + Dexamethasone (N=75)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 0
Diplopia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 3
Hepatitis (Hepatobiliary disorders) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Hepatitis b (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 2 | 1
Genital prolapse (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab + Bortezomib + Dexamethasone (N=75) | Bortezomib + Dexamethasone (N=75)
Anaemia (Blood and lymphatic system disorders) | 25 | 20
Lymphopenia (Blood and lymphatic system disorders) | 5 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 22
Tachycardia (Cardiac disorders) | 3 | 4
Cataract (Eye disorders) | 3 | 4
Vision blurred (Eye disorders) | 4 | 5
Abdominal distension (Gastrointestinal disorders) | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 8
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6
Constipation (Gastrointestinal disorders) | 28 | 21
Diarrhoea (Gastrointestinal disorders) | 31 | 24
Dyspepsia (Gastrointestinal disorders) | 7 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 19 | 16
Vomiting (Gastrointestinal disorders) | 14 | 7
Asthenia (General disorders) | 20 | 21
Chest pain (General disorders) | 6 | 2
Chills (General disorders) | 4 | 2
Face oedema (General disorders) | 4 | 4
Fatigue (General disorders) | 22 | 17
Influenza like illness (General disorders) | 7 | 4
Injection site erythema (General disorders) | 3 | 4
Oedema (General disorders) | 5 | 3
Oedema peripheral (General disorders) | 21 | 18
Pyrexia (General disorders) | 25 | 15
Bronchitis (Infections and infestations) | 8 | 7
Conjunctivitis (Infections and infestations) | 9 | 4
Herpes zoster (Infections and infestations) | 6 | 3
Influenza (Infections and infestations) | 3 | 7
Pneumonia (Infections and infestations) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 10 | 4
Urinary tract infection (Infections and infestations) | 3 | 5
Viral upper respiratory tract infection (Infections and infestations) | 6 | 4
Rib fracture (Injury, poisoning and procedural complications) | 5 | 2
Blood creatinine increased (Investigations) | 5 | 4
Platelet count decreased (Investigations) | 6 | 8
Weight decreased (Investigations) | 7 | 3
Weight increased (Investigations) | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 12 | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 12
Dizziness (Nervous system disorders) | 9 | 7
Dysgeusia (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 8 | 6
Neuralgia (Nervous system disorders) | 5 | 4
Neuropathy peripheral (Nervous system disorders) | 28 | 28
Paraesthesia (Nervous system disorders) | 19 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 9
Somnolence (Nervous system disorders) | 0 | 6
Tremor (Nervous system disorders) | 3 | 5
Anxiety (Psychiatric disorders) | 7 | 2
Confusional state (Psychiatric disorders) | 4 | 2
Depression (Psychiatric disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 20 | 15
Pollakiuria (Renal and urinary disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 8 | 5
Hypertension (Vascular disorders) | 12 | 3
Hypotension (Vascular disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.